CLINICAL TRIAL: NCT04789434
Title: PD-1 Inhibitor Tislelizumab Maintenance Therapy in Newly Diagnosed DLBCL Patients After ASCT: A Multicenter, Randomized Controlled Clinical Study on Efficacy and Safety
Brief Title: PD-1 Inhibitor Tislelizumab Maintenance Therapy in Newly Diagnosed DLBCL Patients After ASCT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Vice President, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NHL-PD1-1
Record Dates: First submitted 2021-03-06; First posted 2021-03-09 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Transplantation; Chemotherapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 Inhibitor maintenance (Experimental): PD-1 Inhibitor Tislelizumab maintenance therapy dose：200mg frequency：1 time for 2 months duration：2 years
  Interventions: Drug: PD-1 Inhibitor Tislelizumab maintenance therapy
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Drug: PD-1 Inhibitor Tislelizumab maintenance therapy — PD-1 Inhibitor Tislelizumab maintenance therapy, 200mg, every 2 months, 12 times
  Arms: PD-1 Inhibitor maintenance

SUMMARY:
This is a multicenter, randomized controlled, prospective clinical trial. The objective is to investigate the efficacy and safety of Tislelizumab maintenance therapy in newly diagnosed diffuse large B-cell lymphoma (DLBCL) patients after autologous hematopoietic stem cell transplantation (ASCT).

DETAILED DESCRIPTION:
This is a multicenter, randomized controlled, prospective clinical trial. The objective is to investigate the efficacy and safety of Tislelizumab maintenance therapy in newly diagnosed diffuse large B-cell lymphoma (DLBCL) patients after autologous hematopoietic stem cell transplantation (ASCT). 94 patients were randomly divided into two groups according to the ratio of 1:1. The whole trial included screening period (day-28 to day-1), treatment period (Tislelizumab, 200mg every 8 weeks, 12 times) and follow-up period (2 years after the enrollment).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female, aged 18-65;
2. newly-diagnosed high risk (aaipi 2-3 and aaipi 1 with large mass) DLBCL patients after autologous stem cell transplantation;
3. Laboratory tests (blood tests, liver and renal function) meet the following requirements:

   1. Blood tests: white blood cell count ≥ 3.0 × 109 / L, absolute neutrophil count ≥ 1.5 × 109 / L, hemoglobin ≥ 90g / L, platelet ≥ 75 × 109 / L
   2. Liver function: transaminase ≤ 2.5 × upper limit of normal value, bilirubin ≤ 1.5 × upper limit of normal value;
   3. Renal function: serum creatinine 44-133 mmol / L;
4. The score of ECOG was 0-2;
5. The subject or his legal representative must provide written informed consent before the special examination or procedure of the study.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Severe complications or infection;
3. Lymphoma involving central nervous system;
4. Participate in other clinical trials at the same time;
5. According to the judgment of the researcher, the patients who are not suitable for this study were selected.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2-years after enrollment
  Progression-free survival was defined as the time from the date of diagnosis until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria,or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
complete remission rate | 2-years after enrollment
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria
overall survival | 2-years after enrollment
  Overall survival was defined as the time from the date of diagnosis to the date of death from any cause. Reported is the percentage of participants with event. of disease progression or relapse, using 2014 Lugano criteria,or death from any cause, whichever occurred first.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No